CLINICAL TRIAL: NCT00285012
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial With 40-Week Follow-Up Evaluating The Safety And Efficacy Of Varenicline Tartrate For Smoking Cessation In Patients With Mild-To-Moderate Chronic Obstructive Pulmonary Disease
Brief Title: Smoking Cessation in Subjects With Mild-to-moderate Chronic Obstructive Pulmonary Disease (COPD).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3051054
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; smoking cessation in COPD
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- varenicline (Experimental)
  Interventions: Drug: Varenicline Tartarate

INTERVENTIONS:
Drug: placebo — 1mg (placebo) by mouth twice daily for 12 weeks (first week is up titration schedule---0.5mg once daily for 3 days, 0.5mg twice daily for 4 days)
  Arms: placebo
Drug: Varenicline Tartarate — 1 mg by mouth twice daily for 12 weeks (first week is up titration schedule---0.5mg once daily for 3 days, 0.5mg twice daily for 4 days)
  Other Names: Chantix, Champix
  Arms: varenicline

SUMMARY:
This study is to be conducted in subjects with mild-to-moderate COPD who are cigarette smokers with the intent of demonstrating differences in smoking cessation between varenicline and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be current cigarette smokers who have smoked an average of at least 10 cigarettes per day during the past year and during the month prior to the screening visit.
* mild to moderate COPD confirmed by spirometry
* Subjects must have a clinical diagnosis of COPD.

Exclusion Criteria:

* Subjects who have made a serious attempt to quit smoking in the past 3 months.
* Subjects who have been previously randomized in a study that has included varenicline.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2006-05; Primary Completion 2008-07 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (18):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Portland, Maine
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
- France (4):
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
- Italy (3):
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Vittorio Veneto, TV
- Spain (3):
  - Pfizer Investigational Site, L'hospitalet Del Llobregat, Barcelona
  - Pfizer Investigational Site, Cáceres, Caceres
  - Pfizer Investigational Site, Madrid, Madrid

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Tashkin DP, Rennard S, Taylor Hays J, Lawrence D, Marton JP, Lee TC. Lung function and respiratory symptoms in a 1-year randomized smoking cessation trial of varenicline in COPD patients. Respir Med. 2011 Nov;105(11):1682-90. doi: 10.1016/j.rmed.2011.04.016. Epub 2011 May 31. PMID 21621992
- [Derived] Tashkin DP, Rennard S, Hays JT, Ma W, Lawrence D, Lee TC. Effects of varenicline on smoking cessation in patients with mild to moderate COPD: a randomized controlled trial. Chest. 2011 Mar;139(3):591-599. doi: 10.1378/chest.10-0865. Epub 2010 Sep 23. PMID 20864613
- [Derived] Ryerson CJ, Berkeley J, Carrieri-Kohlman VL, Pantilat SZ, Landefeld CS, Collard HR. Depression and functional status are strongly associated with dyspnea in interstitial lung disease. Chest. 2011 Mar;139(3):609-616. doi: 10.1378/chest.10-0608. Epub 2010 Aug 5. PMID 20688924
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051054&StudyName=Smoking%20cessation%20in%20subjects%20with%20mild-to-moderate%20Chronic%20Obstructive%20Pulmonary%20Disease%20%28COPD%29.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were current cigarette smokers 35 years of age or older with mild to moderate Chronic Obstructive Pulmonary Disease (COPD) as defined by Global Initiative for Chronic Obstructive Lung Diseases (GOLD) criteria.
Groups:
- Varenicline: Varenicline 0.5 milligrams (mg) once daily (QD) for 3 days; followed by 0.5 mg twice daily (BID) for 4 days; then 1 mg BID for 11 weeks.
- Placebo: Placebo 0.5 milligrams (mg) once daily (QD) for 3 days; followed by 0.5 mg twice daily (BID) for 4 days; then 1 mg BID for 11 weeks.
Period: Assigned to Study Treatment (Tx)
Arm/Group | Varenicline | Placebo
Started | 250 | 254
Completed | 248 | 251
Not Completed | 2 | 3
Not completed — Other | 2 | 3
Period: Received Study Tx
Arm/Group | Varenicline | Placebo
Started | 248 | 251
Completed Tx (May Continue in Study) | 207 (After treatment completion at Wk 12, subjects may continue in nontreatment follow-up phase) | 193 (After treatment completion at Wk 12, subjects may continue in nontreatment follow-up phase)
Discontinued Tx (May Continue in Study) | 41 (Discontinued Tx=12 Adverse Event (AE); 10 Lost to follow up; 13 subject withdrawal; 6 other, unknown) | 58 (Discontinued Tx=14 AE;3 Lack of efficacy;10 Lost to follow up;25 subject withdrawal;6 other, unknown)
Completed | 176 (Completed study through nontreatment follow-up phase Week 13 to Week 52) | 157 (Completed study through nontreatment follow-up phase Week 13 to Week 52)
Not Completed | 72 | 94
Not completed — Death | 2 | 1
Not completed — Adverse Event | 5 | 11
Not completed — Lack of Efficacy | 0 | 3
Not completed — Lost to Follow-up | 29 | 31
Not completed — Withdrawal by Subject | 31 | 43
Not completed — Other | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 248 | 251 | 499
Age Continuous [Mean (Standard Deviation); unit: years] | 57.2 (9.1) | 57.1 (9.0) | 57.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 95 | 188
  Male | 155 | 156 | 311

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Four Week Continuous Quit Rate (CQR)
Description: Number of subjects who reported no smoking and no use of other nicotine-containing products since the last study visit (on the Nicotine Use Inventory [NUI]) and with end-expiratory exhaled carbon monoxide (CO) measurement less than or equal to 10 parts per million (ppm) for weeks 9 through 12 (inclusive).
Time Frame: Week 9 through Week 12
Population: All subjects population: received at least 1 dose, including partial doses, of randomized study drug.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
participants | 105 | 22
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Primary endpoint was based on a CO confirmed 4-week CQR (weeks 4 through 12 inclusive). Intent was to evaluate the alternative hypothesis that varenicline is superior to placebo for smoking cessation after 12 weeks of treatment in subjects with mild to moderate COPD; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 8.40, 95% CI [4.99 to 14.14] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center

2. Secondary Outcome: Number of Subjects With Continuous Abstinence (CA)
Description: Number of subjects who reported no smoking and no use of other nicotine-containing products (treatment phase = through week 12) or tobacco products (non-treatment phase = after treatment phase; follow up through week 52) at each contact (on the NUI) and with end-expiratory exhaled CO measurement less than or equal to 10 ppm from week 9 through week 24 and week 52. CO confirmed in-clinic visit.
Time Frame: Week 9 through Week 24 and Week 52
Population: All subjects population
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
participants
  Week 9 | 125 | 28
  Week 24 | 64 | 18
  Week 52 | 46 | 14
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Varenicline versus (vs) placebo at Week 24; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 4.88, 95% CI [2.75 to 8.65] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 52; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 4.04, 95% CI [2.13 to 7.67] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center

3. Secondary Outcome: Number of Subjects With Long Term Quit Rate (LTQR)
Description: Number of subjects who were responders for the primary endpoint (4-week CQR for Weeks 9 through 12) and who had no more than 6 cumulative days of smoking from Week 12 through the given visit (Week 24 and Week 52).
  CO confirmed in-clinic visit.
Time Frame: Week 24, Week 52
Population: All subjects population
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
participants
  Week 24 | 70 | 19
  Week 52 | 53 | 17
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 24; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 5.17, 95% CI [2.96 to 9.02] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 52; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 3.92, 95% CI [2.18 to 7.07] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center

4. Secondary Outcome: Number of Subjects With 7-Day Point Prevalence of Abstinence
Description: Number of subjects at given visit (Week 12, Week 24, Week 52) or telephone contact, reported no smoking and no use of other nicotine-containing products (treatment phase) or tobacco products (non-treatment phase) in the last 7 days and with end-expiratory exhaled CO measurement less than or equal to 10 ppm. CO confirmed in-clinic visit.
Time Frame: Week 12, Week 24, Week 52
Population: All subjects population
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
participants
  Week 12 | 119 | 31
  Week 24 | 74 | 34
  Week 52 | 65 | 36
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 12; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 6.99, 95% CI [4.39 to 11.11] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 24; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 2.85, 95% CI [1.79 to 4.54] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 52; Test type: Superiority or Other; p = 0.0008, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 2.19, 95% CI [1.37 to 3.48] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center

5. Secondary Outcome: Number of Subjects With 4-Week Point Prevalence of Abstinence
Description: Number of subjects at Week 52 visit reporting no smoking and no use of other tobacco products in the last 4 weeks and with end-expiratory exhaled CO measurement less than or equal to 10 ppm.
Time Frame: Week 52
Population: All subjects population
Measure: Number; unit: particpants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
particpants | 65 | 33
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 52; Test type: Superiority or Other; p = 0.0002, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and pooled center; Odds Ratio (OR) = 2.45, 95% CI [1.52 to 3.95] — odds ratio obtained from a logistic regression model including the main effects of treatment and pooled center

6. Secondary Outcome: Change From Baseline in Pre-bronchodilator and Post-bronchodilator Forced Expiratory Volume in First Second (FEV1)
Description: Change from baseline in mean FEV1 (forced expiratory volume in the first second of forced exhalation) measured in millimeters (ml) as mean at observation minus baseline value. Directly after pre-bronchodilator measurement, subject inhaled albuterol or salbutamol delivered by metered-dose inhaler (MDI); post-bronchodilator lung function repeated 30 to 45 minutes following administration of albuterol or salbutamol.
Time Frame: Baseline, Week 12, Week 52
Population: All subjects population; (n) = subjects with analyzable data at observation for varenicline and placebo, respectively. Missing data imputed by carrying the last observation forward (LOCF), including baseline values.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
ml
  Week 12 [LOCF] Pre-bronchodilator (n= 244, 248) | 33.69 (281.08) | 1.77 (282.28)
  Week 12 [LOCF] Post-bronchodilator (n=237, 246) | 73.84 (287.20) | 15.61 (223.02)
  Week 52 [LOCF] Pre-bronchodilator (n=244, 248) | -29.59 (276.53) | -37.90 (286.47)
  Week 52 [LOCF] Post-bronchodilator (n=237, 246) | -8.10 (285.80) | -9.51 (277.46)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 12 [LOCF] pre-bronchodilator; Test type: Superiority or Other; p = 0.140, ANCOVA; p-value based on ANCOVA model with treatment and center as factors and baseline value as covariate
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 12 [LOCF] post-bronchodilator; Test type: Superiority or Other; p = 0.007, ANCOVA; p-value based on ANCOVA model with treatment and center as factors and baseline value as covariate
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 52 [LOCF] pre-bronchodilator; Test type: Superiority or Other; p = 0.684, ANCOVA; p-value based on ANCOVA model with treatment and center as factors and baseline value as covariate
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Varenicline vs placebo at Week 52 [LOCF] post-bronchodilator; Test type: Superiority or Other; p = 0.901, ANCOVA; p-value based on ANCOVA model with treatment and center as factors and baseline value as covariate

7. Secondary Outcome: Change From Baseline in Clinical COPD Questionnaire (CCQ)
Description: Change from baseline: mean at observation minus baseline value. Subject-administered 10-item instrument to systematically assess COPD symptoms (items 1, 2, 5, and 6), functional states (items 7, 8, 9, and 10) and mental states (items 3 and 4); For each domain score = sum of items divided by the number of items; total score = sum of scores divided by 10; range from 0 (very good health) to 6 (extremely poor health). Assessed at each visit based on subject's experience during the week prior to visit.
Time Frame: Baseline, Week, 12, Week 24, Week 52
Population: All subjects; (n) = subjects with analyzable data at observation for varenicline and placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
scores on scale
  Week 12 Mental State (n=214, 193) | -0.81 (1.25) | -0.64 (1.31)
  Week 24 Mental State (n=191, 161) | -0.72 (1.36) | -0.49 (1.43)
  Week 52 Mental State (n=174, 155) | -0.58 (1.37) | -0.46 (1.39)
  Week 12 Functional State (n=214, 192) | -0.41 (0.98) | -0.35 (1.00)
  Week 24 Functional State (n=191, 160) | -0.40 (1.01) | -0.25 (1.02)
  Week 52 Functional State (n=175, 154) | -0.35 (0.96) | -0.12 (1.06)
  Week 12 Respiratory Symptoms (n=213, 193) | -1.16 (1.19) | -0.88 (1.17)
  Week 24 Respiratory Symptoms (n=191, 161) | -0.98 (1.08) | -0.82 (1.14)
  Week 52 Respiratory Symptoms (n=175, 155) | -0.90 (1.16) | -0.63 (1.36)
  Week 12 Total Score (n=213, 192) | -0.79 (0.91) | -0.62 (0.93)
  Week 24 Total Score (n=191, 160) | -0.70 (0.89) | -0.52 (0.93)
  Week 52 Total Score (n=174, 154) | -0.62 (0.89) | -0.39 (1.05)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Week 12 Mental State; Test type: Superiority or Other; p = 0.078, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Week 24 Mental State; Test type: Superiority or Other; p = 0.109, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Week 52 Mental State; Test type: Superiority or Other; p = 0.281, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 4: Comparison: Varenicline vs Placebo; Week 12 Functional State; Test type: Superiority or Other; p = 0.581, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 5: Comparison: Varenicline vs Placebo; Week 24 Functional State; Test type: Superiority or Other; p = 0.290, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 6: Comparison: Varenicline vs Placebo; Week 52 Functional State; Test type: Superiority or Other; p = 0.063, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 7: Comparison: Varenicline vs Placebo; Week 12 Respiratory Symptoms; Test type: Superiority or Other; p = 0.002, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 8: Comparison: Varenicline vs Placebo; Week 24 Respiratory Symptoms; Test type: Superiority or Other; p = 0.081, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 9: Comparison: Varenicline vs Placebo; Week 52 Respiratory Symptoms; Test type: Superiority or Other; p = 0.016, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 10: Comparison: Varenicline vs Placebo; Week 12 Total Score; Test type: Superiority or Other; p = 0.033, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 11: Comparison: Varenicline vs Placebo; Week 24 Total Score; Test type: Superiority or Other; p = 0.078, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate
Statistical Analysis 12: Comparison: Varenicline vs Placebo; Week 52 Total Score; Test type: Superiority or Other; p = 0.023, ANCOVA; p-value obtained from ANCOVA model with fixed effect terms for center and treatment, and baseline score as a covariate

8. Secondary Outcome: Number of Cigarettes Smoked Daily During First 3 Weeks of the 12-Week Treatment Period
Description: Number of cigarettes smoked daily collected during the first 3 weeks of study after randomization using patient smoking diaries.
Time Frame: Day 1 through Day 21
Population: All subjects population; (n) = number of subjects who smoked at least 1 cigarette at the given day for varenicline and placebo, respectively.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
cigarettes per day
  Day 1 (n=226, 231) | 19.9 (11.0) | 18.7 (9.8)
  Day 2 (n=232, 230) | 18.8 (10.6) | 18.4 (9.7)
  Day 3 (n=233, 233) | 17.7 (9.9) | 17.4 (9.6)
  Day 4 (n=230, 232) | 17.1 (9.7) | 17.1 (9.5)
  Day 5 (n=224, 228) | 16.5 (9.6) | 16.9 (9.3)
  Day 6 (n=222, 230) | 16.4 (9.9) | 16.0 (9.1)
  Day 7 (n=214, 228) | 15.9 (11.3) | 15.3 (9.9)
  Day 8 (n=176, 201) | 13.9 (12.0) | 13.4 (9.9)
  Day 9 (n=168, 193) | 12.2 (9.8) | 12.7 (9.5)
  Day 10 (155, 187) | 12.1 (9.1) | 12.6 (8.9)
  Day 11 (n=151, 190) | 11.6 (8.3) | 12.1 (9.0)
  Day 12 (n=145, 188) | 11.4 (8.5) | 11.9 (8.9)
  Day 13 (n=144, 184) | 11.1 (8.5) | 11.9 (8.9)
  Day 14 (n=134, 183) | 11.1 (8.8) | 12.9 (11.6)
  Day 15 (n=131, 180) | 11.1 (8.5) | 11.5 (8.7)
  Day 16 (n=132, 179) | 10.8 (8.7) | 11.9 (9.2)
  Day 17 (n=128, 176) | 10.5 (8.3) | 11.9 (9.3)
  Day 18 (n=123, 176) | 10.7 (8.3) | 11.9 (9.3)
  Day 19 (n=120, 176) | 10.1 (7.9) | 11.6 (8.7)
  Day 20 (n=121, 162) | 9.7 (8.6) | 11.3 (7.9)
  Day 21 (n=100, 132) | 9.8 (8.8) | 10.4 (8.2)

9. Secondary Outcome: Change From Baseline in Inflammatory Biomarkers: C-Reactive Protein (CRP) and Fibrinogen Antigen
Description: Change from baseline in CRP and Fibrinogen antigen (blood markers of inflammation) calculated as mean at observation minus baseline value; measured as milligrams per deciliter (mg/dl).
Time Frame: Baseline, Week 12, Week 52
Population: All subjects population; (n) = number of subjects with analyzable data at observation for varenicline and placebo, respectively.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 248 | 251
mg/dl
  Week 12 CRP (n=210, 197) | -0.0 (1.0) | -0.0 (1.0)
  Week 52 CRP (n=162, 146) | 0.0 (0.9) | 0.1 (0.8)
  Week 12 Fibrinogen (n=183, 174) | -25.2 (100.6) | -1.4 (86.9)
  Week 52 Fibrinogen (n=150, 130) | -8.2 (102.1) | 14.9 (79.2)

10. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline calculated as mean at observation minus baseline value; body weight measured in kilograms (kg).
Time Frame: Baseline, Week 52
Population: Subjects with change in body weight in the All subjects population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 217 | 205
kg | 2.4 (6.3) | 1.5 (4.0)

ADVERSE EVENTS:
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 6/248 | 11/251
Other Adverse Events (participants affected / at risk) | 157/248 | 121/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=248) | Placebo (N=251)
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=248) | Placebo (N=251)
Abdominal pain (Gastrointestinal disorders) | 7 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 0
Constipation (Gastrointestinal disorders) | 12 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 9
Dry mouth (Gastrointestinal disorders) | 12 | 4
Dyspepsia (Gastrointestinal disorders) | 9 | 1
Flatulence (Gastrointestinal disorders) | 18 | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 67 | 20
Vomiting (Gastrointestinal disorders) | 16 | 6
Fatigue (General disorders) | 11 | 1
Irritability (General disorders) | 6 | 4
Bronchitis (Infections and infestations) | 9 | 11
Influenza (Infections and infestations) | 5 | 3
Nasopharyngitis (Infections and infestations) | 10 | 11
Rhinitis (Infections and infestations) | 6 | 3
Sinusitis (Infections and infestations) | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 22 | 20
Weight increased (Investigations) | 11 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Dizziness (Nervous system disorders) | 4 | 7
Dysgeusia (Nervous system disorders) | 7 | 6
Headache (Nervous system disorders) | 20 | 20
Abnormal dreams (Psychiatric disorders) | 27 | 7
Anxiety (Psychiatric disorders) | 5 | 5
Depression (Psychiatric disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 24 | 15
Nightmare (Psychiatric disorders) | 5 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other